CLINICAL TRIAL: NCT01359423
Title: Comparison of Primary Long Full Coverage Stenting vs Primary Short Spot Stenting for Long Femoropopliteal Artery Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2010-0065
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- long coverage (Experimental): Primary long full coverage stenting
  Interventions: Drug: Percutaneous transluminal angioplasty of femoropopliteal artery lesions with primary long
- short spot (Active Comparator): primary short spot stenting
  Interventions: Drug: short stenting for the primary outcome and use of cilostazol for 12 months for secondary outcome.

INTERVENTIONS:
Drug: Percutaneous transluminal angioplasty of femoropopliteal artery lesions with primary long — Patients will be randomized in a two-by-two factorial manner according to the use of IVUS guidance (IVUS guidance vs. no IVUS guidance) for the PCI and the duration of dual anti-platelet therapy (100 mg/day aspirin and 75mg/day clopidogrel for 6 months vs. 12 months) after PCI. Each randomization of the enrolled subjects will be done 1:1.
  Arms: long coverage
Drug: short stenting for the primary outcome and use of cilostazol for 12 months for secondary outcome. — Patients will be randomized in a two-by-two factorial manner according to the use of IVUS guidance (IVUS guidance vs. no IVUS guidance) for the PCI and the duration of dual anti-platelet therapy (100 mg/day aspirin and 75mg/day clopidogrel for 6 months vs. 12 months) after PCI. Each randomization of the enrolled subjects will be done 1:1.
  Arms: short spot

SUMMARY:
Hypothesis: Primary long full coverage stenting is superior to primary short spot stenting in the treatment of long (≥80 mm) femoropopliteal artery lesions.

Study design :

* Prospective, randomized, multi-center study
* A total of 220 subjects with symptomatic peripheral artery disease of lower limbs who meet all inclusion and exclusion criteria will be included.
* Patients will be randomized in a two by two factorial manner according to the strategy of stenting (long versus short stenting) and the additional use of cilostazol. Each randomization of the enrolled subjects will be done 1:1.
* Patients will be followed clinically for 1 year after the procedure.
* Angiographic or CT follow-up will be performed at 1 year.

ELIGIBILITY:
Inclusion Criteria:

Clinical criteria:

1. Age 20 years of older
2. Symptomatic peripheral artery disease:

   * Moderate or severe claudication (Rutherford category 2 or 3)
   * Critical limb ischemia (Rutherford category 4 or 5)
3. Patients with signed informed consent

Anatomical criteria:

1. Target lesion length ≥80 mm by angiographic estimation
2. Stenosis of more than 50 percent or occlusion of the ipsilateral superficial femoral artery
3. At least one patent (less than 50 percent stenosed) tibioperoneal runoff vessel.

Exclusion Criteria:

Clinical criteria

1. Acute critical limb ischemia
2. Severe critical limb ischemia (Rutherford category 6)
3. Major bleeding history within prior 2 months
4. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel or contrast agents
5. Age > 85 years
6. Severe hepatic dysfunction (> 3 times normal reference values)
7. Significant renal dysfunction (Serum creatinine > 2.0 mg/dl
8. Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
9. LVEF < 40% or clinically overt congestive heart failure
10. Pregnant women or women with potential childbearing
11. Life expectancy <1 year due to comorbidity

Angiographic criteria

1. Previous bypass surgery or stenting of the superficial femoral artery
2. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
The rate of binary restenosis | 12months after the index procedure
  The rate of binary restenosis (stenosis of at least 50 percent of the luminal diameter) in the treated segment 12 months after intervention, as determined by computed tomographic angiography (CTA) or catheter angiography according to the stenting strategy

SECONDARY OUTCOMES:
Ankle-brachial index, etc | at 12 months according to the stenting strategy
  1. Ankle-brachial index at 12 months according to the stenting strategy
  2. Maximal walking distance at 12 months according to the stenting strategy
  3. The rate of reintervention including repeat endovascular therapy or bypass surgery involving the target lesion
  4. The rate of limb salvage at 12 months according to the stenting strategy
  5. The rate of major adverse cardiovascular events (MACE) at 12 months according to the stenting strategy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea